CLINICAL TRIAL: NCT06671678
Title: Long-Term Prognosis Of An Implant Osteointegrated With The Root Remnant On-Site: A Case Report
Brief Title: Dental Implant Osteointegrated With The Residual Root
Status: Active, not recruiting | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esra UYGUÇ, Principal Investigator, Ege University
Other Study IDs: EGE-PRTZ-EU-001
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Dental Implant Failed; Osteointegration; Dental Crowns
Keywords: Root remnant; Dental implant failed; osteointegration; Dentine-implant interface

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This case report presents the long-term prognosis of an implant resulting in late failure with an osteointegrated root remnant on the fixture 11 years after implant placement. A 68-year-old female patient experienced issues with a maxillary right 4-unit implant-supported bridge placed 11 years ago. During removal, an osteointegrated root remnant was discovered on the middle supporting implant, which had been inadvertently placed over it. Clinicians should be cautious with retained root remnants, as they may impact osteointegration. However, both the implant and root fragment were osteointegrated without adverse effects.

DETAILED DESCRIPTION:
There is a growing demand for implant dentistry as the first rehabilitation choice for treating patients with missing teeth. Clinicians can encounter asymptomatic retained root fragments in edentulous spaces. This case report presents the long-term prognosis of an implant resulting in late failure with an osteointegrated root remnant on the fixture 11 years after implant placement. A 68-year-old female patient presented to the clinic with complaints of function related to a maxillary right 4-unit implant-supported bridge 11 years after the first insertion of the implants. After removal of the restoration, a root remnant was observed as osteointegrated on the fixture of the middle supporting implant. The implant was placed encroaching upon the mesial part of the residual root fragment left unintentionally, which was discovered accidentally during bridge removal. Clinicians should show ultimate attention when utilizing the retained root remnants in implant sites considering the potential risk of hindering osteointegration. However, osteointegration of the encroached implant and root fragment is plausible, with no observed adverse effects. A risk-benefit evaluation should be assessed individually.

ELIGIBILITY:
Inclusion Criteria:

* Patient with dental implants placed in contact with residual roots

Exclusion Criteria:

* Lack of retained root remnants
* Lack of dental implants

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with dental implants placed in contact with residual roots
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Dental Implant Osteointegrated With The Residual Root | From enrollment to the end of treatment at 11 years
  The prognosis of the osseointegration status of the retained root remnant and dental implant over an 11-year follow-up period.
  Whether osseointegration has occurred will be verified based on follow-up radiographic images and periodically recorded examination data. Evaluation criteria include implant stability, compatibility with surrounding bone and soft tissues, and potential inflammatory reactions around the root remnant. These measures are intended to understand the long-term integration of the implant and root remnant.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Uyguç, Principal Investigator — Ege University Faculty of Dentistry Department of Prosthodontics
Locations (1):
- Ege University Faculty of Dentistry Department of Prosthodontics, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Uyguc E, Yaylaci E, Koyuncu B, Kumbuloglu O. Implant Osseointegration Adjacent to a Retained Root Fragment: A Case With 11-Year Follow-up. Case Rep Dent. 2025 Jul 20;2025:5547549. doi: 10.1155/crid/5547549. eCollection 2025. PMID 40726544
- See also: Immediate Loading of Implants Inserted Through Impacted Teeth in the Esthetic Area: A Series of 10 Cases with up to 7 Years of Follow-up — https://pubmed.ncbi.nlm.nih.gov/30986281/
- See also: When should root remnants and unrestorable broken teeth be extracted in frail older adults? — https://pubmed.ncbi.nlm.nih.gov/34392937/
- See also: Attachment of Residual Root onto Dental Implant: A Case Report with Literature Review — http://www.ijcpd.org/journal/view.html?volume=15&number=4&spage=226&year=2019